CLINICAL TRIAL: NCT02399306
Title: A Prospective, Multicenter, Randomized Controlled Study to Compare Chemoradiotherapy With or Without Enteral Nutrition Intervention for Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma
Brief Title: Chemoradiotherapy With or Without Enteral Nutrition for Locally Advanced Thoracic Esophageal Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Collaborators: Wuhan University (Other); Xiangya Hospital of Central South University (Other); Shanxi Province Cancer Hospital (Other); Shandong Tumor Hospital (Other); Henan Cancer Hospital (Other Government); Peking University Cancer Hospital & Institute (Other); Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, LI TAO, Section Head, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: scch2015001
Record Dates: First submitted 2015-03-17; First posted 2015-03-26 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Esophageal Squamous Cell Carcinoma; Enteral Nutrition Therapy; Chemoradiotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Enteral Nutrition; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): chemoradiotherapy with Enteral Nutrition intervention
  Interventions: Drug: Enteral nutrition; Radiation: radiotherapy
- Arm B (Placebo Comparator): chemoradiotherapy
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Drug: Enteral nutrition — Patients in the Trial Group received concurrent chemoradiotherapy and standardized, whole-course enteral nutrition management.
  Arms: Arm A
Radiation: radiotherapy — Patients receive intensity modulated radiation therapy(IMRT) from week 1 to week 7,once a day, 5 times per week.
  Radiotherapy dose：95% gross tumor volume（GTV-T） 60-66 Gy /30-33f，GTV-N 60-66 Gy /30-33f，CTV-T 50-54 Gy /25-27f，CTV-N 50-54 Gy /25-27f.

SUMMARY:
This is a randomized, prospective, multicenter study.

DETAILED DESCRIPTION:
This is a randomized, prospective, multicenter study. The aim of this study was to compare the changes of body weight,survival,toxicity,quality of life and opportunistic infection frequency in Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma between and after chemoradiotherapy with or without enteral nutrition therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old
* male or femalePathologically or cytologically proven esophageal squamous cell carcinoma
* Clinical stage II or stage III
* PG-SGA≧2
* Karnofsky performance score(KPS) ≧70
* Estimated life expectancy of at least 12 weeks
* Hemoglobin≥90.0g/dL,white blood cell count（WBC）≥ 4000 cells/mm³,Platelet count≥100,000 cells/mm³
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times upper limit of normal,bilirubin normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Patients have good compliance to treatment and follow-up of acceptance
* Forced expiratory volume in one second（FEV1） ≥ 1.5 litre or ≥ 75% of the reference value
* the functions of the heart, kidney, liver were basically normal, with no chemotherapy and radiotherapy contraindications

Exclusion Criteria:

* Patients with severely bowel function impaired or can not tolerate enteral nutrition
* Patients with serious gastrointestinal obstruction, be unable to take food by mouth and can not / do not want to a feeding tube inserted
* Patients have no risk of malnutrition
* Patients have severe malnutrition (weight loss >10% or <30 g/L, BMI<18.5 kg/m2 or hemoglobin<90 g/L before the treatment
* Patients who have severe vomiting, gastrointestinal bleeding, intestinal obstruction
* Patients can not tolerate chemotherapy and radiotherapy
* Patients who have distant metastasis
* The primary tumor or lymph node already received surgical treatment (except for biopsy);
* Patient who received radiotherapy for primary tumor or lymph node;
* Patient who received chemotherapy or immunotherapy;
* Patient who suffered from other malignant tumor;
* Patient who have taken other drug test within 1 month;
* Pregnant woman or Lactating Women and Women in productive age who refuse to take contraception in observation period;
* Subject with a severe allergic history or idiosyncratic;
* Subject with severe pulmonary and cardiopathic disease history;
* Refuse or incapable to sign the informed consent form of participating this trial;
* Drug abuse or alcohol addicted;
* Subject with a Personality or psychiatric diseases, people with no legal capacity or people with limited capacity for civil conduct;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Body Weight Change from baseline to the end of treatment | up to 1 month after the treatment
  Body weight change from baseline to the end of treatment = body weight at the end of treatment - baseline body weight.

SECONDARY OUTCOMES:
Maximum Body Weight Change during treatment | up to 1 month after the treatment
  Maximum body weight change during treatment= the lowest body weight during treatment - baseline body weight.
Blood biochemical examination | up to 1 month after the treatment
  albumin, haemoglobin,et al
Grade 3-5 toxicity | up to 1 month after the treatment
  Grade 3-5 adverse events as assessed by NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0 andthe criteria of the Radiation Therapy Oncology Group ，such as esophagitis、pneumonitis 、hematologic toxicity and infection rate
Completion rate of chemoradiotherapy | up to 1 month after the treatment
  The proportion of people who complete all treatment as required
short-term effect | up to 1 month after the treatment
  objective remission rate
Overall Survival | at least 2 years
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: TAO LI, MD, PhD, Study Chair — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sichuan Cancer Hospital & Institute, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Lyu J, Shi A, Li T, Li J, Zhao R, Zhu S, Wang J, Xing L, Yang D, Xie C, Shen L, Zhang H, Zhu G, Wang J, Pan W, Li F, Lang J, Shi H. Effects of Enteral Nutrition on Patients With Oesophageal Carcinoma Treated With Concurrent Chemoradiotherapy: A Prospective, Multicentre, Randomised, Controlled Study. Front Oncol. 2022 Feb 25;12:839516. doi: 10.3389/fonc.2022.839516. eCollection 2022. PMID 35280748